CLINICAL TRIAL: NCT02817373
Title: Implantation Prediction Model by the Use of Three Dimensional (3D) Ultrasound in Fresh Embryo Transfers Cycles
Brief Title: Implantation Prediction by Three Dimensional (3D) Ultrasound in Fresh Embryo Transfers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 123-16MMC
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Infertility
Keywords: IVF; embryo transfer; ultrasound; implantation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transvaginal ultrasound study (Other): Patients with a well established infertility requiring IVF treatment and who are <40. Cohort will consist of patients going through a fresh day 5 transfer with a planned transfer of a single good quality embryo. Patients will go thorough a Ultrasound scan performed through a vaginal probe on the morning of the embryo transfer.
  Interventions: Other: Ultrasound scan performed through a vaginal probe

INTERVENTIONS:
Other: Ultrasound scan performed through a vaginal probe — 5-8 minute scan recording : endometrial thickness, endometrial pattern, endometrial -myometrial junction appearance, subendometrial wave contractions (presence and number), endometrial surface area

SUMMARY:
This study is designed to predict implantation of a fresh, high quality embryo in an in vitro fertilization (IVF) cycle by using ultrasound based uterine factors.

DETAILED DESCRIPTION:
Investigators will recruit patients <40 years with no background morbidities who are being treated with IVF or IVF intra cytoplasmic sperm injection (ICSI) for acceptable indications. Only patients reaching a blastocyst transfer will be recruited ; this criterion will assist in minimizing embryonal quality as a factor in the implantation chance. The investigators will limit the quality to good quality embryos, which in the unit's routine practice are transferred in a single embryo transfer. On Day 5, embryos will be scored for blastocyst formation. Blastocysts will be graded according to the size of the blastocyst, the assessment of the inner cell mass (ICM) and trophectoderm development as suggested by Gardner. Good quality embryos (Grade 1-2) will be defined as those where at least: "3" score if the cavity completely fills the embryo, "B" when the ICM is loosely grouped with several cells and "B" when the trophectoderm has very few cells forming a loose epithelium. Lower criteria embryos on Day 5 will be defined as poor quality embryos (Grade 3 or 4). Blastocyst grading will be performed by two trained embryologists, each with over 10 years of experience. The study will not involve any change in the conventional IVF treatment; the only change will involve a 3D trans-vaginal ultrasound at the morning of the embryo transfer, before patients are initiating bladder filling (a common request from all abdominally assisted embryo transfers, facilitating an easier pathway to the uterus and an excellent view). The estimated time for the ultrasound test is 5-8 minutes and will include recording of the following variables : endometrial thickness, endometrial pattern, endometrial -myometrial junction appearance, subendometrial wave contractions (presence and number), endometrial surface area. The information will be recoded under the patients' unique study identity number and will be stored in a special computerized archived file secured by Meir medical center data protection and computer unit. The data will not affect any treatment decisions in the IVF unit unless this examination will reveal for the first time the presence of an unknown uterine polyp or the presence of a hydrosalpinx. Such scenario is improbable since in the performing unit, patients are routinely going through a uterine cavity assessment and a pelvic ultrasound scan prior to an IVF cycle. If this indeed happens then the ultrasound unit will contact the IVF unit and the treating physician will discuss the data with the patient in order to decide whether to go on with the transfer or to freeze the embryo/s until treating the new findings. Upon completion of 150 patients/studies, the ultrasound file will be analyzed by two highly trained and experienced examiners. Each of the variables collected will be used in a multivariate model for implantation incorporating the patient's age.

ELIGIBILITY:
Inclusion Criteria:

* Single day 5 fresh embryo transfer of good quality
* Age<40

Exclusion Criteria:

* Frozen embryo transfer
* Age>40
* Day 2-3 transfer
* Double embryo transfer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
implantation of a fresh high quality embryo | outcome measure will be known within 4 weeks of the embryo transfer
  Implantation is defined as the presence of a gestational sac as will be assessed by a vaginal ultrasound probe 4 weeks after the embryo transfer. Implantation is expected to exist only in cases of a positive pregnancy test; in such cases the ultrasound can either describe an absence of sac, a single sac or multiple sacs.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Wiser, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Result] Matsuura K, Hayashi N, Takiue C, Hirata R, Habara T, Naruse K. Blastocyst quality scoring based on morphologic grading correlates with cell number. Fertil Steril. 2010 Aug;94(3):1135-7. doi: 10.1016/j.fertnstert.2009.11.003. Epub 2010 Jan 15. PMID 20079898
- [Result] Hershko-Klement A, Tepper R. Ultrasound in assisted reproduction: a call to fill the endometrial gap. Fertil Steril. 2016 Jun;105(6):1394-1402.e4. doi: 10.1016/j.fertnstert.2016.04.012. Epub 2016 Apr 29. PMID 27140291